CLINICAL TRIAL: NCT04888169
Title: Optimizing Attention Bias Modification for Posttraumatic Stress Disorder: An Entirely Remote Study
Brief Title: Studying the Modification of Attention Bias Remotely After Trauma
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19-27541
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Attention bias
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (7):
- Attention Bias Modification - Word Stimuli (Experimental): Attention bias modification training involves a probe detection task as follows: (1) a fixation cross appears on the screen for 500ms; (2) the fixation cross is replaced by two target stimuli (one threat word and one neutral word) that are displayed at the top and the bottom of the screen for 500ms; (2) the stimuli disappear and a visual probe appears (the letter E or F), in the location of one of the two stimuli until the participant responds to indicate whether the letter was an E or an F using response buttons at the bottom of the phone screen. In the active ABM condition, the probe replaces the neutral stimulus 100% of the time.
  Interventions: Device: SMART Mobile App - Attention Bias Modification
- Attention Bias Modification - Face Stimuli (Active Comparator): Attention bias modification training involves a probe detection task as follows: (1) a fixation cross appears on the screen for 500ms; (2) the fixation cross is replaced by two target stimuli (one threatening face and one neutral face) that are displayed at the top and the bottom of the screen for 500ms; (2) the stimuli disappear and a visual probe appears (the letter E or F), in the location of one of the two stimuli until the participant responds to indicate whether the letter was an E or an F using response buttons at the bottom of the phone screen. In the active ABM condition, the probe replaces the neutral stimulus 100% of the time.
  Interventions: Device: SMART Mobile App - Attention Bias Modification
- Attention Control Training - Word Stimuli (Experimental): Attention control training involves a probe detection task as follows: (1) a fixation cross appears on the screen for 500ms; (2) the fixation cross is replaced by two target stimuli (i.e. one threat word and one neutral word) that are displayed at the top and the bottom of the screen for 500ms; (2) the stimuli disappear and a visual probe appears (the letter E or F), in the location of one of the two stimuli until the participant responds to indicate whether the letter was an E or an F using response buttons at the bottom of the phone screen. In the active ACT condition, the probe replaces the neutral stimulus 50% of the time, and replaces the threat stimulus the other 50%.
  Interventions: Device: SMART Mobile App - Attention Control Training
- Attention Control Training - Face Stimuli (Active Comparator): Attention control training involves a probe detection task as follows: (1) a fixation cross appears on the screen for 500ms; (2) the fixation cross is replaced by two target stimuli (one threatening face and one neutral face) that are displayed at the top and the bottom of the screen for 500ms; (2) the stimuli disappear and a visual probe appears (the letter E or F), in the location of one of the two stimuli until the participant responds to indicate whether the letter was an E or an F using response buttons at the bottom of the phone screen. In the active ACT condition, the probe replaces the neutral stimulus 50% of the time, and replaces the threat stimulus the other 50%.
  Interventions: Device: SMART Mobile App - Attention Control Training
- Placebo Attention Training - Word Stimuli (Placebo Comparator): Placebo attention training involves a probe detection task as follows: (1) a fixation cross appears on the screen for 500ms; (2) the fixation cross is replaced by two target stimuli (two neutral words) that are displayed at the top and the bottom of the screen for 500ms; (2) the stimuli disappear and a visual probe appears (the letter E or F), in the location of one of the two stimuli until the participant responds to indicate whether the letter was an E or an F using response buttons at the bottom of the phone screen.
  Interventions: Device: SMART Mobile App - Placebo Training
- Placebo Attention Training - Face Stimuli (Placebo Comparator): Placebo attention training involves a probe detection task as follows: (1) a fixation cross appears on the screen for 500ms; (2) the fixation cross is replaced by two target stimuli (two neutral faces) that are displayed at the top and the bottom of the screen for 500ms; (2) the stimuli disappear and a visual probe appears (the letter E or F), in the location of one of the two stimuli until the participant responds to indicate whether the letter was an E or an F using response buttons at the bottom of the phone screen.
  Interventions: Device: SMART Mobile App - Placebo Training
- Control - Questions (Sham Comparator): The Control - Questions condition will only deliver a set of daily questions for participants to answer. Questions will ask about a variety of psychological factors such as mood, stress experiences, daily exercise and more.
  Interventions: Device: SMART Mobile App - Control

INTERVENTIONS:
Device: SMART Mobile App - Attention Bias Modification — ABM involves placing the probe behind the neutral stimulus on 100% of the trials.
  Arms: Attention Bias Modification - Face Stimuli; Attention Bias Modification - Word Stimuli
Device: SMART Mobile App - Attention Control Training — ACT involves placing the probe behind the neutral stimulus on 50% of trials, and behind the threat stimulus on 50% of trials.
  Arms: Attention Control Training - Face Stimuli; Attention Control Training - Word Stimuli
Device: SMART Mobile App - Placebo Training — Placebo training only includes neutral stimuli.
  Arms: Placebo Attention Training - Face Stimuli; Placebo Attention Training - Word Stimuli
Device: SMART Mobile App - Control — Participants will only answer questions.
  Arms: Control - Questions

SUMMARY:
The investigators will complete an entirely remote randomized controlled trial (RCT) comparing 14 sessions of attention bias modification (ABM), attention control training (ACT), placebo neutral attention training, and a final control condition with daily questions in 1,897 individuals with clinically significant Post-traumatic Stress Symptoms (PTSS) (defined as PCL-5 score ≥ 33). To assess effects of the training and control conditions, the investigators will administer tests of threat-related attention bias and variability, and self-report assessments of PTSS, depression, anxiety, and perceived stress at baseline, after one and two weeks of training, and at eight-week follow up. The investigators plan to screen and confirm interest from over 3,000 eligible participants over a period of 24 months to enroll and randomize 1,897 participants with the end goal of 1,232 completers (176 per condition).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* Score at or above 33 on the PCL-5,
* Able and willing to perform daily smartphone training for two weeks
* Fluent English comprehension.
* Owns Android or iPhone smartphone

Exclusion Criteria:

* Does not have Android or iPhone Operating System (iOS) smartphone running sufficient software (i.e. at least iOS 10.1), and is not willing to update
* Active suicidality.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1314 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in PTSD Checklist-5 (PCL) Score (Before/After Training) | Baseline, 4 weeks
  Looking at the change of PCL scores from prior to beginning (baseline) and directly after completing the training at week 4. PCL scores range from 0-80 with a score of 33 indicating clinically significant levels of PTSD. A 10 point change (up or down) is considered a clinically significant change in PTSD symptoms.
  A PCL score of <33 indicates non-clinically significant PTSS. A PCL score of >= 33 indicates clinically significant PTSS.
Change in PTSD Checklist-5 (PCL) Score (Follow-up) | 4 weeks, 8 Weeks
  Looking at the change of PCL scores from directly after completing the training at 4 weeks to a follow-up conducted at week 8. PCL scores range from 0-80 with a score of 33 indicating clinically significant levels of PTSD. A 10 point change (up or down) is considered a clinically significant change in PTSD symptoms.
  A PCL score of <33 indicates non-clinically significant PTSS. A PCL score of >= 33 indicates clinically significant PTSS.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Woolley, MD, PhD, Principal Investigator — UCSF, SFVAMC; Joaquin Anguera, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Tommy Atwater, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No